CLINICAL TRIAL: NCT06460467
Title: Semi-automatic Segmentation Method for Determining 177Lu-DOTATATE Tumor Dosimetry
Acronym: SSTR
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI103
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Meningioma
Keywords: dosimetry; theragnostic
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with 177Lu-DOTATATE: Patients treated with 177Lu-DOTATATE for a meningioma at the Nancy University Hospital and for a neuroencrine tumor in the EVADOVE study NCT04467567 (who underwent scintigraphy on D1, D4 and D7 (± 1 day)
  Interventions: Device: scintigraphy of 177Lu-DOTATATE

INTERVENTIONS:
Device: scintigraphy of 177Lu-DOTATATE — The medical device under study is a hybrid wide-field CZT solid-state camera, the VERITON-CT ™ camera.

SUMMARY:
The aim of this study was to compare a semi-automatic segmentation method with manual reference segmentation to determine an overall tumor volume on post-therapy scintigraphy at D1 in patients treated with 177Lu-DOTATATE for meningioma or neuroendocrine tumor for dosimetric calculation.

DETAILED DESCRIPTION:
The new wide-field solid-state cameras enable "quantitative" single-photon emission tomoscintigraphy (SPECT) acquisitions, particularly during internal vectorized radiotherapy treatments. These innovative treatments are mainly used in cancer therapy. They involve the injection of a radiopharmaceutical consisting of a vector specifically targeting the tumor cell - in this case, somatostatin analogues targeting somatostatin receptors - and a radioactive isotope emitting β- or α-radiation to "kill" the tumor cell, and γ-radiation for SPECT imaging - in this case 177Lu. These radiopharmaceuticals are currently prescribed at fixed doses for all patients. With the aim of personalized medicine, tumor dosimetry is essential for predicting efficacy and dose-response relationships at the individual level of this type of treatment. In view of the increasing therapeutic applications of these 177Lu therapies, the European Association of Nuclear Medicine (EANM) has recently issued recommendations on the dosimetry of 177Lu-labeled somatostatin analogues (Lutathéra®, 177Lu-DOTATATE), among others.

Nevertheless, these recommendations are precise as regards dosimetry to organs at risk, but remain unclear as regards tumor dosimetry. Tumor dosimetry is therefore difficult to implement on a routine clinical basis.

The efficacy of 177Lu-DOTATATE treatment has been demonstrated for neuroendocrine tumors in the NETTER-1 phase 3 study, and interesting results have been reported for the treatment of refractory meningiomas.

Furthermore, a recent study showed that in patients with gastrointestinal neuroendocrine tumors treated with 177Lu-DOTATATE, tumor dosimetry could predict patient survival.

In order to optimize a dosimetric approach in clinical routine, several steps are necessary: i) define a standardized manual or semi-automated segmentation method for determining the volumes of interest (tumor volume and/or organs at risk), ii) precisely quantify tumor or organs at risk volume activities over time, and iii) determine the doses absorbed by the tumor and/or organs at risk.

An initial study was conducted in the department of nuclear medicine,to define a semi-automatic segmentation method for meningiomas treated with 177Lu-DOTATATE on pre-therapeutic 68Ga-DOTATOC positons emission tomography (PET), with the aim of predicting tumor dosimetry from pretherapeutic imaging. For this study, tumor segmentation will be performed directly on SPECT imaging carried out post-treatment on a 360° wide-field CZT camera to determine tumor dosimetry.

The aim of this study is to compare a semi-automatic segmentation method with manual reference segmentation to determine overall tumor volume on post-therapy scintigraphy at D1 in patients treated with 177Lu-DOTATATE for meningioma or neuroendocrine tumor, with a view to dosimetric calculation.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with 177Lu-DOTATATE for meningioma at Nancy University Hospital
* Patients with neuroendocrine tumors in the EVADOV study who underwent scintigraphy on D1, D4 and D7 (± 1 day)

Exclusion Criteria:

* Patients who refused to have their data used retrospectively

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with 177Lu-DOTATATE for a meningioma at Nancy University Hospital and for a neuroendocrine tumor in the EVADOV study who underwent scintigraphy at D1, D4 and D7 (± 1 day)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Dice index | 1 day
  Dice index between semi-automatic segmentation and reference segmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy, France